CLINICAL TRIAL: NCT01162590
Title: Reactogenicity and Safety of a Single Dose of GlaxoSmithKline (GSK) Biologicals' Human Rotavirus (HRV) Vaccine (444563) in Healthy Adults
Brief Title: Study to Evaluate the Reactogenicity and Safety of Rotarix™ in Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113545
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Infections, Rotavirus
Keywords: Human Rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Rotarix Group (Experimental): Subjects will receive Rotarix™.
  Interventions: Biological: Rotarix ™
- Placebo Group (Placebo Comparator): Subjects will receive placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix ™ — Oral, single dose
  Arms: Rotarix Group
Biological: Placebo — Oral, single dose
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the safety of Rotarix ™ when administered in healthy adults aged 18 to 45 years in China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female subject of Chinese origin, 18 years to 45 years inclusive of age at the time of the vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests.
* Any clinically significant history of chronic gastrointestinal disease including uncorrected congenital malformation of gastrointestinal tract that would predispose for Intusussception.
* Gastroenteritis within 7 days preceding the study vaccine or placebo administration.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination. Planned administration/ administration of a vaccine not foreseen by the study protocol within 14 days of the study vaccine or placebo and ending 14 days after.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Administration of immunoglobulins and/ or any blood products within the three months preceding the dose of study vaccine or planned administration during the study period.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/ or drug abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-03-31 (Actual); Study Completion 2010-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of each solicited symptom | Within the 8-day (Day 0 - Day 7) follow-up period after the vaccine dose

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse events | Within 31 days (Day 0 - Day 30) after the vaccine dose
Occurrence of serious adverse events | Throughout the study period following the vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Liucheng County, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Li RC, Li YP, Mo ZJ, Luo D, Huang T, Kong JL, Wang LH, Song NS, Liu A, Zhang H, Liao X, Karkada N, Han HH. Reactogenicity and safety of a liquid human rotavirus vaccine (RIX4414) in healthy adults, children and infants in China: randomized, double-blind, placebo-controlled Phase I studies. Hum Vaccin Immunother. 2013 Aug;9(8):1638-42. doi: 10.4161/hv.25076. Epub 2013 Jun 4. PMID 23807360
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113545 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113545?search=study&b%22b''%22#rs
- Available data/document: Individual Participant Data Set: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register